CLINICAL TRIAL: NCT00963183
Title: A Phase I, Single Centre, Double-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability and Pharmacokinetics of Inhaled AZD5423 After Single Ascending Doses in Healthy Male Subjects
Brief Title: AZD5423 Single Ascending Dose Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: D2340C00001
Record Dates: First submitted 2009-08-17; First posted 2009-08-21 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2014-11

CONDITIONS: Healthy Volunteers
Keywords: Safety; Tolerability; Healthy; Inhalation
MeSH Terms: conditions — Respiratory Aspiration | interventions — 2,2,2-trifluoro-N-(1-((1-(4-fluorophenyl)-1H-indazol-5-yl)oxy)-1-(3-methoxyphenyl)-2-propanyl)acetamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Drug: AZD5423
  Interventions: Drug: AZD5423
- B (Placebo Comparator): Drug: Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD5423 — Solution for nebulisation, inhaled. Each subject will receive a single-dose of AZD5423 or placebo. Starting dose 8.4µg (lung deposited dose) with up to 8 dose escalations not exceeding AstraZeneca pre-defined exposure limits.
  Arms: A
Drug: Placebo — Solution for nebulisation, inhaled. Each subject will receive a single-dose.
  Arms: B

SUMMARY:
The aim of the study is to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of AZD5423 following single ascending dose administrations in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed, written and dated informed consent prior to any study specific procedures
* Have a body mass index (BMI) between 18 and 30 kg/m2 and weigh at least 50 kg and no more than 100 kg

Exclusion Criteria:

* Any clinically significant disease or disorder
* Any clinically significant abnormalities at screening examination
* Use of any prescribed or non-prescribed medication

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2009-08; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Safety variables (ECG, adverse events, blood pressure, pulse, body temp, safety lab), lung function and physical examination | Frequent sampling occasions during study days

SECONDARY OUTCOMES:
Pharmacokinetics - Maximum plasma concentration (Cmax), time to Cmax (tmax), area under the plasma concentration-time curve from zero to the time of the last measurable concentration [AUC(0-t)] and from zero to infinity (AUC) | Frequent sampling occasions during study days
Add'l pharmacokinetics - Terminal rate constant (λz); terminal half-life (t½λz), Apparent plasma clearance (CL/F), apparent volume of distribution during terminal phase (Vz/F), mean residence time (MRT). | Frequent sampling occasions during study days
Pharmacodynamics - Plasma cortisol concentrations | Frequent sampling occasions during study days

CONTACTS AND LOCATIONS:
Overall Officials: Jorup Carin, Study Director — AstraZeneca R&D, Lund, Sweden; Darren Wilbraham, Principal Investigator — Guy's Drug Research Unit, Quintiles Ltd, London, UK
Locations (1):
- Research Site, London, United Kingdom

REFERENCES:
- See also: Study Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1254&filename=Study_Synopsis_D2340C00001.pdf